CLINICAL TRIAL: NCT03648957
Title: Lifestyle Counselling as Secondary Prevention in Patients With Minor Stroke and Transient Ischemic Attack: A Randomized Controlled Feasibility Study
Brief Title: Lifestyle Counselling as Secondary Prevention in Patients With Minor Stroke and Transient Ischemic Attack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Metropolitan University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-17040484
Record Dates: First submitted 2018-08-14; First posted 2018-08-28 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Transient Ischemic Attack
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Ischemic Attack, Transient | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral intervention (Experimental): Usual stroke service care plus additional lifestyle counselling focusing on smoking cessation, physical activity, and adherence to preventive medication. Regular follow-up sessions (3-4 weeks intervals). Physical activity is monitors by an activity tracker.
  Interventions: Behavioral: Lifestyle counselling; Device: Activity tracker
- Usual care (Active Comparator): Usual stroke service care; including computed tomography brain scan, neurological evaluation, and relevant cardiological/vascular evaluation (48-72 hour telemetry, echocardiography, carotic ultrasound imaging). At discharge all patients will receive written and verbal encouragement to a healthy lifestyle.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Lifestyle counselling — First behavioral counselling session will be conducted before discharge and follow-up session will be offered with 3-4 weeks intervals either by telephone or in the outpatient clinic.
  Arms: Behavioral intervention
Behavioral: Usual care — Usual stroke care discharge session; including written and verbal encouragement to a healthy lifestyle.
  Arms: Usual care
Device: Activity tracker — Participants are encouraged to wear a activity tracker to monitor their physical activity
  Arms: Behavioral intervention

SUMMARY:
Interventions to improve health behaviour in patients with resent acute stroke are not well established. This study will evaluate the feasibility and effect of an early initiated counselling intervention targeting smoking, physical activity, and adherence to preventive medication, with regular follow-up sessions, in patients with acute minor stroke or transient ischemic attack who are discharged home.

DETAILED DESCRIPTION:
Stroke is a significant cause of morbidity, mortality, and loss of independence worldwide. In Denmark 12,000 people have a stroke per year. About one fourth of patients admitted with a stroke have had previous strokes or transient ischemic attack (TIA). The risk of recurrent stroke is highest in the first weeks and decreasing with time.

In the last decades there has been an increased focus on the importance of health behaviour in the public and among patients in relations to prevention of vascular diseases. There is solid scientific evidence of the harmful effects of lifestyle factors, such as smoking, physical inactivity, and alcohol overuse.

Hypertension is one of the leading risk factors for vascular diseases, including stroke and TIA. Lowering of the blood pressure is therefore an essential part of stroke treatment. Smoking cessation, physical activity, and adherence to antihypertensive and antithrombotic medication is highly recommended in patients with minor stroke and TIA.

There is still a lack of knowledge about how to support patients in making suitable choices to prevent recurrence and progression of their disease. Previous research has shown varying results and it is therefore difficult to point out any specific intervention or element of interventions which would be feasible to implement in clinical practice.

The hypothesis of the study is that early client-centred patient counselling with repeated follow-up sessions after discharge can reduce the blood pressure through smoking cessation, physical activity, and improved adherence to preventive medication in patients with minor stroke and transient ischemic attacks compared to simple encouragement to lifestyle change.

The overall purpose of our research is to develop effective and clinically feasible interventions to prevent recurrent strokes in patients with minor stroke and transient ischemic attacks, and identify unmet needs in the newly discharged patients and their relatives.

The PhD study will comprise of 1) a randomized feasibility trial (n=40) aiming to test a combined behavioural and clinical intervention with follow-up sessions post-discharge with 3-4 weeks intervals in 12 weeks on reducing blood pressure in patients with minor stroke and transient ischemic attack 2) a qualitative study to explore the patients attitudes and experiences towards medicine adherence, lifestyle changes, social support, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years old
* Hospitalized patients with TIA (ICD-10 G45.9) or stroke (ICD-10 I61, I63, I64) with a Scandinavian Stroke Scale of 45-58. Diagnosis must by confirmed by a neurologist
* Discharge to their own home
* Able to give a valid written consent

Exclusion Criteria:

* Severe barriers to communication
* Not able to use a telephone
* Severe disability prior to the stroke (WHO Performance Status >2; mobilised less than 50 % of the day)
* Requiring specialized rehabilitation
* Active abuse of alcohol or narcotics
* Severe psychiatric illness (affective disease, dementia, schizophrenia, anxiety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | At baseline (0 weeks) and end of intervention (12 weeks)
  Change in resting systolic blood pressure from baseline to three months follow-up

SECONDARY OUTCOMES:
Recruitment rate | 12 weeks
  Proportion of eligible patients included in the study
Adherence rate | From baseline (0 weeks) until the end of intervention (12 weeks)
  Proportion of included participants adhering to and completing the study protocol

OTHER OUTCOMES:
Tobacco smoking (Daily/weekly/rarely/has quit smoking/never smoked) | At baseline (0 weeks) and end of intervention (12 weeks)
  Number of participants currently smoking tobacco (self-reported)
Physical activity (Self-reported time used on light/moderate/strenuous activity or exercise per week) | From baseline (0 weeks) until the end of intervention (12 weeks)
  Time used per week on physical activity (self-reported)
Adherence to preventive medication | Previous seven days until the end of the intervention (12 weeks)
  Proportion of taken/missed doses of preventive medication within the last seven days; antithrombotic, anticoagulants, antihypertensiva & lipid-lowering drugs (self-reported)
Waist/hip ratio | At baseline (0 weeks) and end of intervention (12 weeks)
  Ratio between waist- and hip circumference (cm)
Body mass index | At baseline (0 weeks) and end of intervention (12 weeks)
  Body weight relative to height
Fatigue (Fatigue Assessment Scale) | At the end of the intervention (12 weeks)
  10 item questionnaire with 5-level likert scales assessing health related fatigue and the impact of fatigue on everyday activity
Self-reported health | At baseline (0 weeks) and end of intervention (12 weeks)
  Two item questionnaire
Incidence of vascular events | 52 weeks
  Incidence of new stroke, TIA, ischemic heart disease, or all-cause death (combined)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Christensen, MD, Study Director — Department of Neurology, Nordsjællands Hospital
Locations (1):
- Department of neurology, Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liljehult J, Molsted S, Moller T, Overgaard D, Christensen T. Lifestyle counselling as secondary prevention in patients with minor stroke or transient ischemic attack: a randomized controlled pilot study. Pilot Feasibility Stud. 2024 Mar 22;10(1):50. doi: 10.1186/s40814-024-01478-4. PMID 38519983
- [Derived] Liljehult J, Molsted S, Moller T, Overgaard D, Adamsen L, Jarden M, Christensen T. Lifestyle counselling as secondary prevention in patients with minor stroke and transient ischemic attack: study protocol for a randomized controlled pilot study. Pilot Feasibility Stud. 2020 Mar 25;6:40. doi: 10.1186/s40814-020-00583-4. eCollection 2020. PMID 32226634

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03648957/Prot_SAP_000.pdf